CLINICAL TRIAL: NCT06685393
Title: Effects of Injectable Platelet-rich Fibrin and Platelet-Rich Plasma in Treatment of Diabetic Patients with Stage Ⅱ Grade C Periodontitis (Clinical and Microbiological Study).
Brief Title: Efficacy of Injectable Platelet-rich Fibrin Versus Platelet-Rich Plasma As Adjunctive to Scaling and Root Planning in Non-surgical Periodontal Therapy of Periodontitis Patients
Acronym: PRP-IPRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ELsabbahy Ahmed Mohamed Youssef (Other)
Responsible Party: Sponsor-Investigator, ELsabbahy Ahmed Mohamed Youssef, B.D.S, Faculty of dentistry, Mansoura University 2001. principal Investigator., Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A11060722
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Peridontal Disease
Keywords: periodontitis, PRP, I-PRF
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double (participant, outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group (I) (nondiabetic PRPgroup) (Active Comparator): Group (Ⅰ) (non-diabetic patients): n=10 subdivided into Test side: received scaling and rootplanning plus the subgingival application of PRP.
  Control side: received scaling and rootplanning only.
  Interventions: Procedure: Platelet rich plasma (PRP)
- Group (Ⅱ) (non-diabetic patients): (Active Comparator): Group (Ⅱ) (non-diabetic patients): n=10 subdivided into Test side: received MD plus subgingival application of I-PRF. Control side: received MD only.
  Interventions: Procedure: INJECTABLE PLATELET RICH FIBRIN(I-PRF)
- Group (Ⅲ) (diabetic patients) (Active Comparator): Group (Ⅲ) (diabetic patients): n=10 subdivided into Test side: received MD plus subgingival application of PRP. Control side: received MD only.
  Interventions: Procedure: Platelet rich plasma (PRP)
- Group(Ⅳ) (diabetic patients) (Active Comparator): Group(Ⅳ) (diabetic patients): n=10 subdivided into Test side: received MD plus the subgingival application of I-PRF Control side: received MD only.
  Interventions: Procedure: INJECTABLE PLATELET RICH FIBRIN(I-PRF)

INTERVENTIONS:
Procedure: Platelet rich plasma (PRP) — At the 1st visit, each quadrant is scaled and root planned using an ultrasonic scaler and manual instruments until tactile sensation detects smooth crown and root surfaces these procedures were repeated on both sides starting from 1st visit of treatment,2nd,4th, and 6th-week intervals local anesthetic was utilized in some instances where it was the necessary and subgingival application of (PRP) at test side only at baseline,3ed, 6th week.
  Arms: Group (I) (nondiabetic PRPgroup); Group (Ⅲ) (diabetic patients)
Procedure: INJECTABLE PLATELET RICH FIBRIN(I-PRF) — At the 1st visit, each quadrant is scaled and root planned using an ultrasonic scaler and manual instruments until tactile sensation detects smooth crown and root surfaces these procedures were repeated on both sides starting from 1st visit of treatment,2nd,4th, and 6th-week intervals local anesthetic was utilized in some instances where it was the necessary and subgingival application of (I-PRF) at test side only at baseline,3ed, 6th week.
  Arms: Group (Ⅱ) (non-diabetic patients):; Group(Ⅳ) (diabetic patients)

SUMMARY:
The study aims to evaluate the Efficacy of Injectable Platelet-rich Fibrin versus Platelet-Rich Plasma as adjunctive to scaling and root planning in non-surgical periodontal therapy of Periodontitis patients (Randomized controlled clinical trial)

DETAILED DESCRIPTION:
Mechanical Debridement (MD) is the gold standard procedure for managing periodontal diseases and infection control. Currently, a minimally invasive approach involving using of local platelets concentrates in the treatment of periodontitis, Platelets are nonnuclear secretory cells deduced from bone marrow as protein-producing cells. Upon activation, the platelets produce secretory grains and synthesize proteins. Platelets contain a variety of protein molecules ranging from membrane proteins, cytokines, regulatory proteins, and bioactive peptides.

Platelet-rich plasma (PRP) Is a 1st-generation platelet concentrate containing a high attention of platelet but a minimal amount of natural fibrinogen. The α granules release growth factors in 3-5 days of platelet activation, which sustain their stimulation of the proliferative phase for ten days after release.

Platelet-rich fibrin (PRF) is a second-generation platelet concentrate that was introduced by Choukroun et al. in 2001, It is allowed that PRF can improve tissue regeneration due to its effects on vascularization, capturing the circulating stem cells, immune control, and closure of the epithelium, Injectable PRF (I-PRF) is the liquid form of PRF. I-PRF is a bioactive agent attained by low-speed centrifugation, and it can stimulate tissue regeneration. I-PRF at high concentrations may stimulate the secretion of several growth factors and trigger fibroblast migration. I-PRF is generally used in regenerative treatments, but it has good issues.

Platelet concentrates (PCs) are characterized by an increased level of platelets, which are considered cells with a multifunctional role in antimicrobial host defense. First, platelets give a rapid response to microbial colonization of vascular endothelium and are the earliest cells at the affected site. Platelets can incorporate microbes themselves and perform pathogen clearance, killing or damaging microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* • Participants: Adult healthy individuals between 25-45 years old with no gender predilection diagnosed with periodontitis.

  * Fasting blood sugar (80-100mg/dl): This is the recommended range for non-diabetic patients and is according to the American Diabetes Association.
  * (Hemoglobin A1C (HbA1c) levels recommended by the American Diabetes Association. Patients with an HbA1c level equal to or less than 7% were considered patients with well-controlled DM.
  * Patients with at least two quadrants with pocket depth up to 5 mm.

Exclusion Criteria:

* history of any preceding oral infections or periodontal treatment for at least three months before starting the study.
* Smokers and alcoholic patients
* pregnant, post-menopausal, and lactating women.
* Patients with poor systemic health like uncontrolled diabetes, hypertension, osteoporosis, and collagen disorders are also excluded with
* patients who were on or expected to take antibiotics or anti-inflammatory drugs within the duration of the study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
clinical measurement of plaque index (PI). | 3 months
  It assesses oral hygiene and is based on the recording of soft debris on the teeth, plaque was scored using the plaque indices the Tarski et al Modified Quigley Hein Plaque Index (TQHPI). With the TQHPI, mesial, distal, and mid surfaces of facial and lingual aspects were scored:
  0 = no plaque/debris
  1. = separate flecks of plaque at the cervical margin of the tooth.
  2. = a thin continuous band of plaque (up to 1 mm) at the cervical margin of the tooth.
  3. = a band of plaque wider than 1 mm but covering less than one-third of the crown of the tooth.
  4. = plaque covering at least one-third but less than two-thirds of the crown of the tooth.
  5. = plaque covering two-thirds or more of the crown of the tooth. The index for the tooth was calculated by adding the scores from the six surfaces of the tooth and dividing them by six. For each patient, a plaque index was calculated by adding up the indices for each of the teeth examined and dividing by the number of these teeth.
clinical measurement of sulcular bleeding index (SBI). | 3 months
  In 1971, Muhlemann & Son introduced the SBI, which was defined as follows:
  Score 0 gingiva of normal texture and color, no bleeding. Score 1: gingiva normal, bleeding on probing. Score 2: bleeding on probing, change in color, no edema. Score 3: bleeding on probing change in color, slight oedema. Score 4: either: (a) bleeding on probing, change in color, obvious edema or (b) bleeding on probing, obvious edema.
  Score 5: bleeding on probing and spontaneous bleeding, change in color, marked edema.
clinical measurement of Probing depth (PD). | 3 months
  For all groups, the pocket depth measurement was calculated from the gingival margin to the base of the pocket in each quadrant between the first premolar and 1ST molar. It was taken at 6 locations which were mesiofacial, midfacial, distofacial, mesiolingual, midlingual, and distolingual.
  To the closest millimeter, the standard William's graded probe was employed. It was inserted parallel to the tooth's long axis with light force; if present, any heavy calculus deposits interfering with measurement were removed.
  The measurements were put together before being divided by six to determine the mean value of every tooth.
  Following that, the pocket depth value for each patient was calculated by summing the values of all teeth, and then the total number of teeth tested divided by the sum.
clinical measurement of Clinical attachment level (CAL). | 3 months
  For all groups, in each quadrant CAL is measured from the first premolar to the 2nd molar(in mm). By recording six values for every tooth and dividing them by six, the mean value for each tooth was determined. Then, by dividing the total number of teeth inspected by the sum of teeth, we got the mean value of CAL for each patient. If the CEJ landmark is missing because it has been destroyed by dental caries or has been removed by placement of a dental restoration, another fixed reference point can be used to measure attachment loss. Such landmarks might include the apical margin of a restoration or the incisal edge of a tooth. When attachment loss measurements are taken from a fixed landmark other than the CEJ they are called relative attachment loss measurements. Clinical attachment loss or relative attachment loss measurements are the best way to assess the presence or absence of additional periodontal damage

SECONDARY OUTCOMES:
MICROBIOLOGICAL PARAMETERS | 3 months
  Both periodontal pathogens Porphyromonas gingivalis (Pg) and Prevotella intermedia (PI) were detected within subgingival dental plaque samples at baseline before treatment, 6th, and 12th weeks by semiquantitative culture technique, and the resulting bacteria were identified using (PCR).• Quantification of each organism was done by counting the number of colonies forming units (CFU) on each plate. Because dilutions are based on 1 paper point, the plate count times the dilution factor yielded the total number of organisms per paper point A significant reduction was considered when the CFU/paper point decreased to ≤103; a non-significant reduction was considered when the CFU/paper point was 103-105; and a failure of treatment was considered when the CFU/paper point remained ≥105.

CONTACTS AND LOCATIONS:
Overall Officials: Elsabbahy Ahmed Mohamed youssef, B.D.S, Principal Investigator — Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided